CLINICAL TRIAL: NCT02217956
Title: Phase I Study of Cisplatin Hyperthermic Intraperitoneal Chemotherapy Dose Escalation After Surgery in Patients With Unresectable Stage IIIC Ovarian, Tube or Peritoneal Primary Adenocarcinoma Previously Treated by Chemotherapy and Completed by Bevacizumab for 15 Months
Brief Title: Dose Escalation of Cisplatin Hyperthermic Intraperitoneal Chemotherapy After Surgery in Patients With Unresectable Stage IIIC Ovarian, Tube or Peritoneal Primary Adenocarcinoma
Acronym: CHIPASTIN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-024361-51; 2010/1699 (Other: CSET number)
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Ovarian Adenocarcinoma; Fallopian Tube Adenocarcinoma; Primary Peritoneal Carcinoma
MeSH Terms: interventions — Cisplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HCIP + bevacizumab (Experimental): 4 dose level of cisplatin are planned: Level 1 : 50 mg/m2 (start level) Level 2 : 60 mg/m2 Level 3 : 70 mg/m2 Level 4 : 80 mg/m2 Level -1: 40 mg/m2 (in case of DLT at level 1)
  bevacizumab: Treatment starts between week 10 and 14 after HCIP. Dosage: 15 mg/kg for a total of 22 injections every 3 weeks for 15 months
  Interventions: Drug: Cisplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Cisplatin
Drug: Bevacizumab

SUMMARY:
HCIP has shown efficacy in treatment of peritoneal carcinosis from colorectal background. Few studies have been published on the use of HCIP in peritoneal carcinosis from ovarian background but most of them were non-randomized phase II studies on a small population using different type of drugs and dosage. before this heterogeneity it seems necessary to standardize the utilization modalities of HCIP in peritoneal carcinosis from ovarian background

ELIGIBILITY:
Inclusion Criteria:

1. Stage IIIC unresectable ovarian, tubes or peritoneal primitive adenocarcinoma according to FIGO classification previously treated with 6 cycles of carboplatin-cisplatin neoadjuvant chemotherapy with a response allowing complete surgery after the 6 cycles
2. Time frame between the sixth platin injection and the CRS + HCIP < 10 weeks
3. No disease progression during the neoadjuvant chemotherapy
4. 18 </= âge </= 65 ans
5. Performance Status OMS < 2
6. Hematological function : PNN >/= 1.5x10^9/L, platelets >/= 150x10^9/L, hemoglobin > 9 g /dl (transfusion allowed)
7. Hepatic function : Bilirubin </= 1,5 x LSN, ASAT (SGOT) and ALAT (SGPT) </= 3 x LSN, Phosphatases alkaline </= 3 x LSN
8. No kidney related pathology, plasmatic creatinine < 140 µmol/l, creatinine clearance > 60 ml/min (Cockcroft formula) and urinary strip <2 (If urinary strip >/= 2, proteinuria < 1g/24h)
9. Plasmatic albumine > 25 g/l
10. HIV negative status
11. Affiliation to social security
12. Signed informed consent

Exclusion Criteria:

1. Incomplete cell kill surgery
2. Non-epithelial ovarian cancer
3. Borderline tumors
4. Non in complete remission previous cancer for more than 5 five years before inclusion
5. Uncontrolled high blood pressure (blood pressure > 150/100 mm Hg despite antihypertensive treatment)
6. Previous abdominal or pelvic radiotherapy
7. Previous pathology of the central nervous system, except for well controlled pathology like epilepsy
8. Previous stroke, transient ischemic attacks or subarachnoid hemorrhage
9. Previous pulmonary embolism
10. Pregnant or breastfeeding women (Women in age must have a blood negative pregnancy test at least 15 days before going under surgery)
11. Participation to an other clinical trial within 30 days before inclusion in the study
12. Known hypersensitivity to platin or bevacizumab
13. Not healed wound, ulcer or bone fracture
14. Previous haemorrhagic or thrombotic malfunction < 6 months
15. Significant CArdiovascular disorder including:

    * Heart attack or unstable angina within the 6 months before inclusion
    * Grade > 1 congestive heart failure according to the NYHA classification
    * Uncontrolled cardiac arrhythmia despite of treatment (patients with atrial fibrillation for which the pace is under control can be include)
16. Long term or recent (within 10 days before inclusion) medication using Aspirin at dosage > 325 mg/day
17. Long term or recent (within 10 days before inclusion) medication using anticoagulant per os or parenteral or thrombolytic given at full dosage for therapeutic purpose.
18. Grade > 1 previous sensory and motor neuropathies according to CTC AE V4.0
19. Previous abdominal fistula, GI perforation or intra-abdominal abscess within 6 months before first administration of bevacizumab
20. Proof of any other disease, metabolic malfunction, physical or laboratory exam showing any possibility of disease or condition contraindicating administration of the drug under trial or exsposing the patient to several complications related to the treatment.
21. Persons deprived of liberty
22. Impossibility to comply with the medical following of the treatment for geographical, social or mental reason

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Toxicity | Assessed at week 4 and 8 after HCIP then every 3 weeks up to 15 months
  Using NCI CTCV4

SECONDARY OUTCOMES:
Progression Free Survival | Assessed every 3 weeks from HCIP until progression up to 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France